CLINICAL TRIAL: NCT04944550
Title: Development of New Models for the Evaluation of Preclinical Treatment for Urothelial Carcinomas of the Upper Excretory Tract.
Brief Title: New Models for the Evaluation of Preclinical Treatment for Urothelial Carcinomas of the Upper Excretory Tract.
Acronym: CICLOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: INSERM U1194, Institut de Recherche en Cancérologie de Montpellier, Campus Val d'Aurelle, 34298 Montpellier cedex 5 (Unknown)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2020-2/NH01
Record Dates: First submitted 2021-06-22; First posted 2021-06-29 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Upper Urinary Tract Urothelial Carcinoma; Nephroureterectomy; Tumor; Xenograft Model
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Tumor samples removed by nephroureterctomy will be evaluated at Nîmes University Hospital's Pathological Anatomy and Cytology Department. Part of the tumors are dissected into 2-3 mm3 fragments and quickly transported in cold Roswell Park Memorial Institute medium or a phosphate-buffered saline environment to the animal lab for subcutaneous grafting on mice or to the "Resistance to innovative treatments and therapies" team for soft cell dissociation. Cell suspensions will then be transported on ice to our collaborators at Inovotion Laboratories for grafting into the chorioallantoid membrane of chicken embryos, or used for cold in vitro culture at the animal lab for subcutaneous grafts (patient-derived xenograft models).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Upper Urinary Tract Urothelial Carcinomas are rare, aggressive tumors, accounting for 5 to 10% of all urothelial tumors. These include tumors which develop in the renal cavities (renal pelvis, calices) and ureteral tumors. Nephro-ureterectomy is the standard treatment but 80% of patients will have a relapse within 2 years. Only one trial has (Birtle et al. 2020), has shown the interest of postoperative chemotherapy. Neoadjuvant systemic treatment seems particularly interesting for a population which is going to undergo a nephronic loss and therefore reduction in kidney function which is likely to make patients ineligible for cisplatin. In favor of additional immunotherapy, it has been described that upper excretory tract tumors have a high immunogenic potential with a high rate of microsatellite instability.

From surgical samples of patient tumors obtained after nephroureterectomy or biopsy material collected before treatment, we are going to generate patient-derived cell lines and xenograft models in the mouse. A recent publication has demonstrated the feasibility of this approach by specifying that the capture rate of tumor cells is 50% for patient-derived xenografts and 25% for patient-derived cells (Coleman et al. 2020). As tumors harvested from biopsies do not grow in patient-derived xenografts,we plan to graft the biopsies onto chorioallantoic chicken embryo membranes, a model which has never been used for this indication and which is one of the original features of our approach. These three concomitant approaches will allow us to increase our chances of obtaining stable upper urinary tract urothelial carcinoma lines to be used for the screening and identification of new treatments or new combinations of molecules that would benefit patients with upper urinary tract urothelial carcinomas, knowing that very few studies dedicated to this type of cancer have been conducted or published due to the rarity of the disease and the lack of existing models published on the subject of these particular tumors.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated consecutively at the Urology Andrology Department of Nîmes University Hospital for high grade carcinoma of the pelvis or renal ureter with an indication for total nephroureterectomy decided during a multidisciplinary meeting.
* Patient with a diagnosis of high-grade urothelial carcinoma of the pelvis or renal ureter confirmed by histology (biopsy, biopsy of the ureteroscopic) or by cytology with the presence of :
* High-grade disease on ureteroscopic biopsy OR ;
* High grade disease on urinary cytology AND infiltrating appearance of the renal pelvic wall / ureter on the scanner (the presence of hydronephrosis will be considered as pervasive by definition) with a negative cytoscopy.

Exclusion Criteria:

* Any patient who has undergone previous systemic treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients treated consecutively at the Urology Andrology department of Nîmes University Hospital for high-grade carcinomas of the pelvis or renal ureter for whom a total nephroureterectomy has been indicated during a multidisciplinary meeting. The tumor samples used for our study come from specimens removed surgically. Patients must not have undergone any prior systemic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Histological characteristics of patient-derived xenograft models after staining. | 1-6 months after harvesting
  Microscopic observation of cells after staining with hematoxylin and eosin
Study of genomes of tumor specimens | 1-6 months after harvesting
  Exome sequencing of DNA cells isolated from original patient tumor specimens.
Alterations in the genomes of patient-derived xenograft tumor models | 1-6 months after harvesting
  Exome sequencing of DNA cells isolated from patient-derived xenograft tumor models.
Alterations in the genomes of patient-derived cell line models | 1-6 months after harvesting
  Exome sequencing of DNA cells isolated from patient-derived cell line models.
Study of the transcriptome of patient tumor specimens. | 1-6 months after harvesting
  RNA-sequencing of cells isolated from patient tumor specimens.
Transcriptome of the patient-derived xenograft tumor models. | 1-6 months after harvesting
  RNA-sequencing of cells isolated from patient-derived xenograft tumor models.
Transcriptome of the patient-derived cell line models. | 1-6 months after harvesting
  RNA-sequencing of cells isolated from patient-derived cell line models.

SECONDARY OUTCOMES:
Sensitivity to Cisplatin: patient-derived cell line models | 6-8 months after harvesting
  The MIC 50 test (Minimum Inhibitory Concentration required for cell growth to be inhibited by 50%) will be used in vitro to test the tumor cells' response to Cisplatin.
Sensitivity to Carboplatin: patient-derived cell line models | 6-8 months after harvesting
  The MIC 50 test (Minimum Inhibitory Concentration required for cell growth to be inhibited by 50%) will be used in vitro to test the tumor cells' response to Carboplatin.
Sensitivity to Oxaliplatin: patient-derived cell line models | 6-8 months after harvesting
  The MIC 50 test (Minimum Inhibitory Concentration required for cell growth to be inhibited by 50%) will be used in vitro to test the tumor cells' response to Oxaliplatin.
Sensitivity to Gemcitabin: patient-derived cell line models | 6-8 months after harvesting
  The MIC 50 test (Minimum Inhibitory Concentration required for cell growth to be inhibited by 50%) will be used in vitro to test the tumor cells' response to Gemcitabin.
Tumor size in non-treated patient-derived xenograft models | 1-6 months after harvesting
  The volume of tumors will be measured in mm3.
Sensitivity to Cisplatin: tumor size in treated patient-derived xenograft models | 6-8 months after harvesting
  To test the tumor cells' response to Cisplatin in xenograft models, the volume of tumors will be measured in mm3 and compared with the volume of tumors in the non-treated control group.
Sensitivity to Cisplatin: tumor growth rate in patient-derived xenograft models | 6-8 months after harvesting
  To test the tumor cells' response to Cisplatin in xenograft models, the Tumor Growth Inhibition index, which is defined as (1 - (mean volume of treated tumors)/(mean volume of control tumors)) × 100% will be used.
Sensitivity to Carboplatin: tumor size in treated patient-derived xenograft models | 6-8 months after harvesting
  To test the tumor cells' response to Carboplatin in xenograft models, the volume of tumors will be measured in mm3 and compared with the volume of tumors in the non-treated control group.
Sensitivity to Carboplatin: tumor growth rate in treated patient-derived xenograft models | 6-8 months after harvesting
  To test the tumor cells' response to Carboplatin in xenograft models, the Tumor Growth Inhibition index, which is defined as (1 - (mean volume of treated tumors)/(mean volume of control tumors)) × 100% will be used.
Sensitivity to Oxiplatin: tumor size in treated patient-derived xenograft models | 6-8 months after harvesting
  To test the tumor cells' response to Oxiplatin in xenograft models, the volume of tumors will be measured in mm and compared with the volume of tumors in the non-treated control group.
Sensitivity to Oxiplatin: tumor growth rate in treated patient-derived xenograft models | 6-8 months after harvesting
  To test the tumor cells' response to Oxiplatin in xenograft models, the Tumor Growth Inhibition index, which is defined as (1 - (mean volume of treated tumors)/(mean volume of control tumors)) × 100% will be used.
Sensitivity to Gemcitabine: tumor size in treated patient-derived xenograft models | 6-8 months after harvesting
  To test the tumor cells' response to Gemcitabine in xenograft models, the tumor volume will be measured in mm3 and compared with the volume of tumors in the non-treated control group.
Sensitivity to Gemcitabin: tumor growth rate in treated patient-derived xenograft models | 6-8 months after harvesting
  To test the tumor cells' response to Gemcitabin in xenograft models, the Tumor Growth Inhibition index, which is defined as (1 - (mean volume of treated tumors)/(mean volume of control tumors)) × 100% will be used.

OTHER OUTCOMES:
Patients' gender | Day 0
  The sex of patients will be recorded at the inclusion as Male/Female/Transgender
Patients' age | Day 0
  The age of patients will be recorded at the inclusion in years
Primitive tumor site | Day 0
  The site of the patient's primitive tumor will be recorded at the inclusion
Infiltrative tumor | Day 0
  The tumor will be noted as infiltrative or not (YES/NO) at the inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine HOUEDE, Pr., Principal Investigator — CHU de Nimes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France

REFERENCES:
- [Background] Birtle A, Johnson M, Chester J, Jones R, Dolling D, Bryan RT, Harris C, Winterbottom A, Blacker A, Catto JWF, Chakraborti P, Donovan JL, Elliott PA, French A, Jagdev S, Jenkins B, Keeley FX Jr, Kockelbergh R, Powles T, Wagstaff J, Wilson C, Todd R, Lewis R, Hall E. Adjuvant chemotherapy in upper tract urothelial carcinoma (the POUT trial): a phase 3, open-label, randomised controlled trial. Lancet. 2020 Apr 18;395(10232):1268-1277. doi: 10.1016/S0140-6736(20)30415-3. Epub 2020 Mar 5. PMID 32145825